CLINICAL TRIAL: NCT00000937
Title: Study and Treatment of Post Lyme Disease (STOP-LD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DMID 96-182; R01AI031561-04A1 (NIH)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2005-11

CONDITIONS: Lyme Disease
MeSH Terms: conditions — Lyme Disease | interventions — Anti-Bacterial Agents

INTERVENTIONS:
Drug: Antibiotics

SUMMARY:
The purpose of this study is to see how well antibiotics work in reducing chronic fatigue symptoms, such as tiredness, in patients that were treated for Lyme Disease. Fatigue is a common symptom of Lyme Disease. When fatigue does not improve after treatment, patients are considered to have Post Lyme Syndrome (PLS). The chronic fatigue seen in these patients appears to be related to the initial infection which causes Lyme Disease. It is believed, but not proven, that treatment with antibiotics may be effective in relieving chronic fatigue in PLS patients.

DETAILED DESCRIPTION:
You will be assigned randomly (like tossing a coin) to receive either antibiotics or a placebo (sugar pill). Neither you nor your doctor will know which you are receiving. You will learn to give yourself the injection, and you will remain on your study drug for 28 days. A home health care nurse will visit you twice a week to check the injection site, and at weeks 1 and 3 the nurse will draw blood for laboratory tests. At months 1 and 6, you will be examined to see if you have fewer chronic fatigue symptoms after the antibiotics. This will include a fatigue questionnaire, a test of your mental processing speed, and a test of your cerebrospinal fluid.

ELIGIBILITY:
Inclusion Criteria:

You may be eligible for this study if you:

* Are between 18 and 65 years of age.
* Are a resident of Long Island or greater NY metropolitan area.
* Are fluent in English.
* Have a history of Lyme Disease.
* Have completed antibiotic treatment for Lyme Disease 6 or more months before starting the study.
* Have severe fatigue.
* Are not pregnant or planning to be pregnant.

Exclusion Criteria:

You will not be eligible for this study if you:

* Have or have had major medical, neurologic, or psychiatric disorder.
* Have had prior chronic pain, fatigue, or recurrent severe headaches before the onset of Lyme Disease.
* Have had Fibromyalgia Syndrome.
* Have a history of sleep apnea, narcolepsy, or other serious sleep disorder.
* Have a learning disability.
* Have had head trauma requiring hospitalization.
* Have symptomatic gallbladder disease.
* Are anemic.
* Abuse alcohol or illicit drugs.
* Have been treated with another antimicrobial agent for Lyme Disease within 6 months of study.
* Need to be receiving systemic steroid therapy during drug administration and follow-up.
* Have used benzodiazepines within 1 month of study entry.
* Are allergic to Beta lactams (a class of antibiotics).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55
Dates: Study Completion 2005-11

CONTACTS AND LOCATIONS:
Locations (1):
- Lauren Krupp, Stony Brook, New York, United States